CLINICAL TRIAL: NCT07093710
Title: The Safety and Efficacy of Golidocitinib Combined With Mitoxantrone Hydrochloride Liposome or Chidamide in the Treatment of Relapsed or Refractory Peripheral T-cell Lymphoma: A Prospective, Multicenter, Open-label, Phase Ib/II Clinical Study
Brief Title: Golidocitinib Combined With Mitoxantrone Hydrochloride Liposome or Chidamide in the Treatment of Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, MD. PhD., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-346
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-07

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golidocitinib Combined with Mitoxantrone Hydrochloride Liposome or GemOx (Experimental): In Cohort 1, patients will receive 150mg of Golidocitinib, orally once daily (qd), in combination with Mitoxantrone Hydrochloride Liposome, with an initial dose of 15mg/m² of Liposomal Mitoxantrone. Two dose groups are designed: 15mg/m² and 18mg/m². Each treatment cycle is 28 days. The Mitoxantrone Hydrochloride Liposome injection will be combined with Golidocitinib(150mg, qd) at the RP2D dose level for an extension study.
  In Cohort 2, patients will receive 150mg of Golidocitinib, orally once daily (qd), in combination with Chidamide, with an initial dose of 20 mg (biw) of Chidamide. Two dose groups are designed: 20 mg and 30 mg. Each treatment cycle is 28 days. The Chidamide will be combined with Golidocitinib (150mg, qd) at the RP2D dose level for an extension study.
  Interventions: Drug: Golidocitinib; Drug: Mitoxantrone Hydrochloride Liposome; Drug: Chidamide

INTERVENTIONS:
Drug: Golidocitinib — 150mg, po, qd;
Drug: Mitoxantrone Hydrochloride Liposome — Cohort 1: 15 mg/m2, IV, D1 and 18 mg/m2, IV, D1 (phase Ib); RP2D (II study)
Drug: Chidamide — Cohort 2: Chidamide：20mg/30mg, po, Biw (phase Ib); RP2D (phase II study)

SUMMARY:
This is a prospective, multicenter, open-label, phase Ib/II clinical study to evaluate the safety and efficacy of golidocitinib combined with mitoxantrone hydrochloride liposome or chidamide in the treatment of relapsed or refractory peripheral T-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study; fully understand and be informed about the study and sign the Informed Consent Form (ICF); willing to comply with and capable of completing all trial procedures;
* Diagnosed with PTCL according to the 2022 revised WHO lymphoma classification standards based on pathological diagnosis by the research center
* Using the Lugano 2014 lymphoma efficacy evaluation criteria, the patient must have at least one measurable or evaluable lesion
* Age ≥ 18 years
* Expected survival greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ and bone marrow function

Exclusion Criteria:

* Accompanied by hemophagocytic lymphohistiocytosis (HLH)
* Lymphoma involvement in the central nervous system or meninges
* Active infections
* Uncontrolled clinical cardiac symptoms or diseases
* Currently using (or unable to stop at least one week prior to the first dose) a known CYP3A strong inducer or strong inhibitor.
* Currently using vitamin K antagonists, antiplatelet drugs, anticoagulants (or unable to stop them within one week prior to the start of the study treatment).
* History of Human Immunodeficiency Virus (HIV) infection and/or Acquired Immunodeficiency Syndrome (AIDS).
* Patients with mental disorders or those unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(ORR) for Phase 2 | Up to 24 months
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) as the best response.
Maximum tolerated dose (MTD) for Phase 1b | The first cycle after administration
  To identify the MTD

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to 24 months
  Defined as the proportion of patients who achieve complete remission as the best response
Duration of Response(DOR) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Progression-free survival(PFS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Overall survival(OS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided